CLINICAL TRIAL: NCT04052724
Title: Internet-based Treatment for Informal Caregivers in Lithuania LINGI: a Randomized Control Trial
Brief Title: Internet-based Treatment for Informal Caregivers in Lithuania LINGI
Acronym: LINGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Vilnius University (Other); University of Groningen (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Principal Investigator, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LINGI
Record Dates: First submitted 2019-06-06; First posted 2019-08-12 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Caregiver Distress
Keywords: informal caregivers; internet-based cognitive behaviour therapy; culturally adapted psychotherapy; eHealth; caregiver burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either control or intervention group. Participants in the control group will receive the same treatment once the intervention group is finished with the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group LINGI (Experimental): Trans-diagnostic, 8 module, 8 week long internet intervention for reducing informal caregiver burden
  Interventions: Behavioral: Intervention group LINGI
- Control group (No Intervention): Participants in the control group will be instructed to wait. Once intervention group will be finished, participants in control group will be able to access the same intervention

INTERVENTIONS:
Behavioral: Intervention group LINGI — Intervention based on cognitive behavioural therapy principles and culturally adapted to Lithuanian population. Intervention's main purpose is to reduce caregiver burden and increase quality of life. Intervention contains psycho-educational elements as well as examples and exercises.
  Arms: Intervention group LINGI

SUMMARY:
The purpose of this study is to evaluate efficacy of internet intervention for informal caregivers in Lithuania in reducing their care-giving burden.

DETAILED DESCRIPTION:
Intervention is going to take a form of an Internet based Cognitive Behavioural Treatment program (ICBT) consisting of eight modules. These are the themes, as listed chronologically: Introduction, Thoughts, Stress and relaxation, Problem Solving, Communication, Anxiety, Behavioural Activation, Maintenance. These themes were chosen after considering topics which might be the most useful for someone in a role of an informal caregiver, considering the trans-diagnostic nature of the intervention.

Effect of the intervention will be compared against a wait-list control group. Intervention is in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years old or over
* fluent in comprehending, writing and reading Lithuanian language
* score 24 or more points on the Caregiver Burden Inventory
* spent at least last couple of months for providing care
* must have internet access and ability to use computer or any other compatible device

Exclusion Criteria:

* adverse life experiences as identified by LEC
* alcohol addiction
* having severe physical or mental impairments
* suicide risk
* severe interpersonal violence
* the person in need of care has life expectancy below or approximately around 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change on Caregiver Burden Inventory (CBI) | Pre-treatment, week 4, week 8 and 12 months post-treatment
  This measure is used to evaluate caregiver burden. CBI contains 24 questions that are distributed within 5 facets - Time Dependency, Emotional Health, Development, Physical Health and Social Relationships. Answer options are presented on a 5-item Likert scale and ranges from from 0 ('Never') to 4 ('Nearly Always'). Total score on CBI is summed up and ranges from 0 to 96, higher score indicating higher levels of burden experienced.

SECONDARY OUTCOMES:
Change on Perceived stress scale (PSS-14) | Pre-treatment, week 8 and 12 months post-treatment
  Measure will be used to evaluate levels of experienced stress. It contains 14 questions on a Likert scale ranging from 0 ('Never') to 4 ('Very Often'). Higher score indicates more severe symptoms.
Change on The Patient Health Questionnaire (PHQ-9) | Pre-treatment, week 4, week 8 and 12 months post-treatment
  Measure will be used to evaluate depressive symptoms. It contains 9 questions that must be responded to by choosing an answer from 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
Change on Generalized anxiety disorder (GAD-7) | Pre-treatment, week 4, week 8 and 12 months post-treatment
  Measure will be used to evaluate caregiver anxiety. GAD-7 contains 7 questions that must be responded to by choosing an answer from 4-item Likert scale, where number 0 indicates 'Not at all' and 3 - 'Nearly every day'. Higher score indicates more severe symptoms.
Change on World Health Organisation (WHO-5) | Pre-treatment, week 8 and 12 months post-treatment
  This questionnaire contains 5 statements regarding individual's well-being. Each of the statements must be evaluated using 6-item Likert scale with a score of 0 indicating 'At no time' while a score of 5 - 'All the time'. Higher score indicates higher well-being.
Change on The Brunnsviken Brief Quality of Life Scale (BBQ) | Pre-treatment, week 8 and 12 months post-treatment
  BBQ will be used for evaluating overall quality of life. It contains 12 statements ranging on a Likert scale from 0 - 'Strongly Disagree to 4 - 'Strongly Agree'. Higher score indicates higher quality of life.

OTHER OUTCOMES:
Life Events Checklist (LEC) | Pre-treatment
  This measure will be used for screening for potentially traumatic events in respondent's lifetime. This questionnaire contains 16 questions and a box for mentioning any other stressful events experienced by an individual. There are 6 answer options for: 'Happened to me', 'Witnessed it', 'Learned about it', 'Part of my job', 'Not sure' and 'Doesn't apply'.
The Alcohol Use Disorders Identification Test (AUDIT) | Pre-treatment
  AUDIT will be used for assessing caregiver's alcohol consumption. It contains 10 questions in relation to the alcohol intake. Each question has varying answer options. Higher score indicates higher alcohol consumption and risks associated with it.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biliunaite I, Kazlauskas E, Sanderman R, Truskauskaite-Kuneviciene I, Dumarkaite A, Andersson G. Internet-Based Cognitive Behavioral Therapy for Informal Caregivers: Randomized Controlled Pilot Trial. J Med Internet Res. 2021 Apr 7;23(4):e21466. doi: 10.2196/21466. PMID 33825687